CLINICAL TRIAL: NCT06527690
Title: Race Impact on Efficacy of Niraparib Plus Abiraterone Acetate and Prednisone in Patients With Homologous Repair Deficient Castration-resistant Prostate Cancer
Acronym: REPRESENTATION
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study aimed to include multiple countries in Latin America, but only Brazil was feasible, making the intended ethnic and racial design unviable. Activities were closed and no sites were opened for recruitment.
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 1223; 67652000PCR2006 (Other Grant/Funding Number: Janssen)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Castrate Resistant Prostate Cancer; Homologous Recombination Deficiency
MeSH Terms: conditions — Prostatic Neoplasms | interventions — niraparib; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- self-identified as from Black racial origin irrespective of ethnicity (Experimental): Cohort A will include participants self-identified as from Black origin as defined as having origins in any of the Black racial groups of Africa, as per the FDA Guidance on Collection of Race and Ethnicity Data in Clinical Trials, and irrespective of ethnicity. This includes participants with more than one race, including pardos.
  Interventions: Drug: Niraparib/Abirate rone acetate fixed-dose combination; Drug: Prednisone
- Racially self-identified as Native Indigenous American or self-identified Latino and racially White (Experimental): Cohort B will include participants of the following racial and ethnic backgrounds:
  1. self-identified as from Native Indigenous American origins as per the FDA Guidance on Collection of Race and Ethnicity Data in Clinical Trials, irrespective of ethnicity (this includes participants with more than one race, including mestizos)
  2. self-identified as from White origin as per the FDA Guidance on Collection of Race and Ethnicity Data in Clinical Trials, and ethnically self-identified as Latinos. This includes participants with mixed (or mestizo) races.
  Interventions: Drug: Niraparib/Abirate rone acetate fixed-dose combination; Drug: Prednisone

INTERVENTIONS:
Drug: Niraparib/Abirate rone acetate fixed-dose combination — Participants will receive niraparib/abiraterone acetate fixed-dose combination 100/500 mg 2 tablets once daily on days 1-28 of each 28-day cycle.
Drug: Prednisone — Participants will receive prednisone 5mg 2 tablets once daily on days 1-28 of each 28-day cycle.

SUMMARY:
This is an open-label, multicenter, interventional study in racially self-identified black or ethnically self-identified hispanic and racially self-identified white or native American participants with metastatic castration-resistant prostate cancer whose tumors demonstrate molecular alterations compatible with homologous repair deficiency.

DETAILED DESCRIPTION:
This study will enroll up to 70 participants, divided into two cohorts of 35 each. Cohort A will include participants self-identified as of black origin, as defined by the FDA Guidance on Collection of Race and Ethnicity Data in Clinical Trials, including those with more than one race, such as pardos. Cohort B will include (1) participants self-identified from Native Indigenous American origins and (2) participants self-identified from White origin who ethnically identify as Latinos, both as per the FDA guidance. The study will consist of five phases: Prescreening for biomarker evaluation, Screening, Treatment, Extension, and Follow-Up. Participants will be assessed during prescreening using the sponsor's required assays or previous results from CLIA-certified labs showing a pathogenic germline or somatic HRR alteration.

The combination of niraparib/AA plus prednisone is FDA-approved for treating homologous repair deficient metastatic castration-resistant prostate cancer (HRD mCRPC). Given the benefits of this combination and the lack of representation in previous studies, a placebo-controlled study is deemed unethical. Thus, the study design includes two independent cohorts, both receiving the standard of care treatment. This study aims to provide additional information on the benefits of this therapy in underrepresented populations. Conducted with input from experts in racial inequities, the study results may be shared with participants through a plain language summary. Participants will be fully informed about the study's risks and requirements and will receive new information affecting their participation decision. Consent to participate is voluntary and can be withdrawn at any time without penalty. Written consent will be obtained following regulations and participant preferences.

ELIGIBILITY:
Eligibility criteria - Prescreening Inclusion

Age:

≥18 years of age (or the local legal age of consent)

Participant Origin:

Participants of the following origins:

- COHORT A: Participants self-identified as with black origin as defined as having origins in any of the black racial groups of Africa, as per the FDA Guidance on Collection of Race and Ethnicity Data in Clinical Trials, and irrespective of ethnicity. This includes participants with more than one race, including pardos.

- COHORT B: Participants self-identified from Native Indigenous American origins as per the FDA Guidance on Collection of Race and Ethnicity Data in Clinical Trials, irrespective of ethnicity. This includes participants with more than one race, including mestizos.

OR

- Participants self-identified from White origin as per the FDA Guidance on Collection of Race and Ethnicity Data in Clinical Trials, and ethnically self-identified as Latinos.

Participant and Disease Characteristics

* ECOG Performance Status 0-1
* Histologically or cytologically confirmed metastatic prostate adenocarcinoma
* Metastatic disease documented by conventional imaging with CT or MRI (for soft tissue lesions) or 99mTc bone scan (for bone lesions)

  1. Participants with a single bone lesion on 99mTc bone scan with no other non-nodal metastatic disease must have confirmation of bone metastasis by CT or MRI.
  2. Participants with lymph node-only disease are not eligible.
* Willing to provide tumor tissue (archival) for determination of deleterious germline or somatic HRR gene alterations, if no local (testing done at investigator center or commercial testing) or prior sponsor-approved test result is available.

  1.Testing must demonstrate pathogenic gene alterations in ≥1 of the following genes to proceed to screening: ATM, BRCA1, BRCA2, BRIP1, CDK12, CHEK2, FANCA, HDAC2, or PALB2.
* Castration-resistant disease, defined by the PCWG3 as any of the following criteria while on castrate levels of testosterone (less than or equal to 50 ng/dL):

  1. Visceral Progression OR
  2. Bone progression (2 or more new prostate-cancer related new lesions compared to baseline) OR
  3. PSA Progression, as defined by an increase in two consecutive measurements that fulfills all the following criteria:

     1. The evaluations were performed with a minimum interval of 1 week.
     2. Progressive worsening with an increase of at least 50% compared to baseline.
     3. The minimum value of PSA is ≥ 1 ng/ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
12-month radiographic Progression-Free Survival (rPFS) | 12 months
  Assessed by modified RECIST v1.1 and PCWG3 criteria, and defined as time from enrollment until progression of soft tissue lesions measured by CT or MRI as defined in RECIST 1.1, progression of bone lesions observed by bone scan and based on PCWG3, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cotait Maluf, Principal Investigator — Latin American Cooperative Oncology Group

IPD SHARING:
Plan to Share IPD: Undecided